CLINICAL TRIAL: NCT01677780
Title: A Multi-Center, Open-Label, Extension Study of RO5045337 (MDM2 Antagonist) Administered Orally in Patients Treated With RO5045337 on Previous Roche-Sponsored Phase 1 Cancer Studies
Brief Title: An Extension Study of RO5045337 in Participants Participating in Previous Roche-sponsored Cancer Studies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP28366; 2012-001303-20 (EudraCT Number)
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Myelogenous Leukemia, Chronic, Neoplasms, Myelogenous Leukemia, Acute
MeSH Terms: conditions — Leukemia, Myeloid; Bronchiolitis Obliterans Syndrome; Neoplasms | interventions — RO6839921

ARMS (1):
- RO5045337 (Experimental): Participants will continue the most similar dose and formulation available (which does not exceed the MTD or the maximum safely administered dose for that formulation during Phase 1) and the same schedule of RO5045337 treatment that they were receiving at the time of transitioning from their respective parent clinical study protocols: NO21279 (NCT00623870), NO21280 (NCT00559533), NP25299 (NCT01164033), NP28021 (NCT01605526) or NP28023 (NCT01635296).
  Interventions: Drug: RO5045337

INTERVENTIONS:
Drug: RO5045337 — Participants will receive RO5045337 orally in doses ranging from 20 milligram per square meter (mg/m^2) to 1800 mg/m^2 daily, and up to 1500 mg dose twice daily on a variety of schedules including daily for up to 20 days and weekly dosing for 3 weeks in 28 day cycles until disease progression or unacceptable toxicity with maximum treatment duration of 24 months.
  Other Names: MDM2 ANTAGONIST

SUMMARY:
This open-label, extension study is designed to provide continuing treatment with RO5045337 to participants who have completed parent studies NO21279 (NCT00623870), NO21280 (NCT00559533), NP25299 (NCT01164033), NP28021 (NCT01605526) or NP28023 (NCT01635296). Participants are eligible to participate in this study if they have completed required Phase 1 study assessments for primary objectives of respective parent protocol and are having evidence of clinical benefit (as defined by the parent protocol). Participants will continue the most similar dose and formulation available (which does not exceed the maximum tolerated dose [MTD] or the maximum safely administered dose for that formulation during Phase 1) and the same schedule of RO5045337 treatment that they were receiving at the time of transitioning from the parent clinical study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the inclusion criteria outlined in the respective parent protocols: NO21279 (NCT00623870), NO21280 (NCT00559533), NP25299 (NCT01164033), NP28021 (NCT01605526) or NP28023 (NCT01635296)
* Participants must have completed one of the following clinical study protocols and have been determined to have clinical benefit on treatment at the conclusion of required study analyses as defined in the respective parent protocols: NO21279 (NCT00623870), NO21280 (NCT00559533), NP25299 (NCT01164033), NP28021 (NCT01605526) or NP28023 (NCT01635296)

Exclusion Criteria:

* Participants must meet the exclusion criteria outlined in the respective parent protocols: NO21279 (NCT00623870), NO21280 (NCT00559533), NP25299 (NCT01164033), NP28021 (NCT01605526) or NP28023 (NCT01635296)
* Participants who developed disease progression/ requiring other anti-tumor therapy while in the parent protocol
* Participants who have stopped study drug dosing for greater than 56 days
* Participants continuing to require dose modifications
* Participants with worsening adverse events
* Participants with unrelated adverse events, medical illnesses, or changes in performance status that, per investigator discretion, put them at high risk for continuing participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (3):
  - Sarcoma Oncology Center, Santa Monica, California
  - M.D Anderson Cancer Center; Oncology, Houston, Texas
  - Cancer Therapy & Research Ctr; Dept Institute for Drug Development, San Antonio, Texas
- Princess Margaret Hospital, Medical Oncology & Haematology, Toronto, Ontario, Canada
- Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse, France